CLINICAL TRIAL: NCT03842150
Title: Development and Validation of a Screening Score for the Biliary Atresia in Infantile Cholestasis: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-19-001
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2021-01

CONDITIONS: Biliary Atresia; Neonatal Cholestasis; Infantile Hepatitis Syndrome
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- derivation cohort
  Interventions: Diagnostic Test: biliary atresia screen score
- validation cohort
  Interventions: Diagnostic Test: biliary atresia screen score

INTERVENTIONS:
Diagnostic Test: biliary atresia screen score — The investigators aim to develop a scoring system according to clinical, laboratory, imaging features of biliary atresia in the derivation dataset and tested in the validation datasets.

SUMMARY:
Better survival and prognosis of biliary atresia (BA) depend on early diagnosis and timely Kasai portoenterostomy. Identifying BA from other causes of infantile cholestasis at early stage of the disease still remains a major challenge. In this study, the investigators aim to develop and validate a scoring system to screen BA in infants with cholestasis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of neonatal cholestasis Age at first visit less than 90 days after birth

Exclusion Criteria:

Severe congenital malformation Subjects with missing data

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants with cholestasis inclduing biliary atresia
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and Validation a Screening Score for the biliary atresia in infantile cholestasis | 1 weeks
  Developed a scoring system according to clinical, laboratory, imaging features of BA and test it in the clinical work. The score system might including clay stool, γ-glutamyl transpeptadase, the results of ultrasound and subscales selected for logistic regression. The total score would sum all the subscales up.The investigators grade the patients with the cholestasis screen score to identify patients with biliary atresia. Patients with score ≤ 15 points considered to be the low-risk group, and patients with risk score > 15 points considered the high-risk group, and the score model has no maximum or minimum value.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to share all the individual participant data information available to our cooperative hospitals through emails